CLINICAL TRIAL: NCT01728831
Title: Observational Study of Cerebral Tissue Oxygen Saturation During Blood Transfusion in Severe Traumatic Brain Injured Patients
Brief Title: Study of Cerebral Tissue Oxygenation During Transfusion in Traumatic Brain Injury
Acronym: NIRSTBI
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 11-294
Record Dates: First submitted 2012-11-04; First posted 2012-11-20 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: TBI (Traumatic Brain Injury); Acute Brain Injuries
Keywords: Red Cell Transfusion; Cerebral tissue oxygenation; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This proposal aims to provide some objective, non-invasively achieved, physiologically relevant data in order to provide some rational basis for decision-making for transfusion in sTBI. Specifically this proposal is an observational study of transfusion and brain tissue saturation in sTBI patients. The results will illustrate to what degree brain tissue oxygenation is critically dependent on the degree of anemia in sTBI and help in the decision of whether transfusion might be helpful.

DETAILED DESCRIPTION:
While there are studies that have invasively monitored cerebral saturation and brain tissue oxygen in severe traumatic brain injury (sTBI) patients, there are none using non-invasive cerebral saturation monitoring in TBI patients undergoing packed red blood cell (pRBC) transfusion. To date, all published studies have involved invasive monitoring with their concomitant potential side effects. Insertion of invasive probes and monitors has several risks and side effects including bleeding, local trauma and brain damage, and infection. Furthermore, they have limited utility as information is restricted to the region of the brain surrounding the probe, as opposed to a more global picture. We therefore propose an observational study using non-invasive near infrared spectroscopy to monitor brain tissue oxygen during the transfusion of packed red blood cells.

Primary Hypothesis:

• Improved oxygen delivery causes improved brain tissue oxygen saturation.

Testable Hypothesis:

• The transfusion of packed red blood cells resulting in a change in the hemoglobin in the 70- 100g/L range, will be associated with an increase in cerebral tissue oxygen saturation measured by near infrared spectroscopy in severe traumatic brain injured patients.

Primary Aims:

• Evaluate the applicability of a 4 wavelength near-infrared spectroscopy (NIRS) to monitor the cerebral oximetry in traumatic brain injury patients. Observe the trend of cerebral tissue oxygenation saturations (StO2) before, during and after a blood transfusion in TBI patients.

Secondary Hypothesis:

* We hypothesize that as pRBCs are transfused there will be a plateau (i.e. hemoglobin threshold) beyond which no increase in cerebral tissue oxygenation will occur.
* There will be lag time between the increase in systemic hemoglobin and the improvement of cerebral tissue oxygenation.

Secondary Aims:

* To correlate the systemic hemoglobin level with cerebral tissue oxygenation saturation as pRBCs are transfused.
* Correlation of non-invasive cerebral tissue oxygenation saturation measurements with invasive brain tissue oxygen tension (if available).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patient with clinical diagnosis of severe TBI and GCS <9
3. Patient requiring PRBC transfusion with a qualifying Hb< 10/dL

Exclusion Criteria:

1. Inability to place the NIRS probes on the patients (facial fractures, facial laceration, etc.).
2. Deficient signal of SctO2 impeding its proper valuation
3. Active coronary ischemia as judged by dynamic ischemic ECG changes and/ or positive troponin levels not due to myocardial contusion.
4. Active hemorrhage: Example

   1. Bleeding into the chest, abdomen or retro-peritoneum likely to require surgery +/- embolization
   2. Pelvic fracture likely to require surgery +/- embolization
   3. More than two long bone fractures requiring operative fixation
5. Clinical diagnosis of drug or alcohol intoxication as predominant cause of coma
6. Systolic BP <90mmHg
7. Heart rate > 120bpm
8. GCS=3 + un-reactive pupils

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 Patient with clinical diagnosis of severe TBI and GCS <9 and Age > 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Applicability of a 4 wavelength near-infrared spectroscopy (NIRS) to monitor the CHANGE in absolute cerebral oximetry over time | Compare the change from the start of the transfusion until 10 hours later.
  After the physician in charge for the patient decides a PRBC transfusion is needed, the FORE-SIGHT probe will be placed on the patient's forehead. A single PRBC unit will be transfused over 30 - 60 minutes. Recording will be started 60 minutes before the transfusion and continued for up to 10 hours after the PRBC unit.

SECONDARY OUTCOMES:
The impact of PRBC transfusion on absolute cerebral oximetry compared to peripheral values over time. | Level of hemoglobin and hematocrit on admission, before transfusion and hourly after the transfusion for up to 5 hours
  Blood specimens (2-4 ml each every 30-60 minutes up to 5 hours) will be drawn concurrently with the routine blood work ordered by the clinical team. The additional blood work will be drawn from an arterial line or central line already in place so no needles will be used, thus minimizing the risk further.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Baker, MD, Study Director — Medical Director, Critical Care; Victoria A McCredie, MBChB, Principal Investigator — Sunnybrook Health Sciences Center, University of Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada